CLINICAL TRIAL: NCT02191956
Title: Technology to Enhance Treatment for Early Conduct Problems in Low Income Families
Acronym: TE-HNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0078; R01MH100377 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-07-16 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Disruptive Behavior Disorders
Keywords: Disruptive behavior disorders; Early Onset; Young Children; Parenting; Behavioral Parent Training
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Parent Training (Active Comparator): Standard of care intervention
  Interventions: Behavioral: Behavioral Parent Training
- Behavioral Parent Training - Enhanced (Experimental): Standard of Care Behavioral Parent Training plus new delivery methods
  Interventions: Behavioral: Behavioral Parent Training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — Weekly clinic session, mid-week call, home practice
  Other Names: Parent Management Training

SUMMARY:
This study aims to the test the efficacy and cost effectiveness of new service delivery methods to enhance the reach and impact of the standard of care treatment, Behavioral Parent Training (BPT), for early onset disruptive behavior disorders.

DETAILED DESCRIPTION:
Families will be randomized to one of two active treatment conditions, the standard BPT program or the standard BPT program plus some new service delivery methods.

ELIGIBILITY:
Inclusion Criteria:

* Child aged 3 to 7 years
* has clinically significant disruptive behaviors
* low-income family

Exclusion Criteria:

* Caregiver has current mood, substance use, and/or psychotic disorder
* Child has current pervasive developmental and/or psychotic disorder
* Family has current allegation and/or past substantiation with child protective services

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2013-04; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Engagement | Participants will be followed for the duration of treatment, an expected average of 10 weeks
  Engagement includes multiple dimensions of participation in the treatment process, including items assessing attendance at weekly sessions, participation in mid-week calls, and home practice of skills.

SECONDARY OUTCOMES:
Change in Disruptive Behavior from the start of treatment through 6 months after treatment ends | Participants will be followed through the duration of treatment and 6 additional months after treatment ends, an expected average of 9 months
  Disruptive behavior includes multiple dimensions of behavior, including items assessing noncompliance, aggression, and oppositionality.
Treatment Cost | Treatment costs will be tracked through the duration of treatment, an expected average of 10 weeks
  Cost is a multidimensional measure that includes items assessing both start-up (e.g., technology development) and implementation (e.g., therapist time) costs.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Jones, Ph.D., Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Department of Psychology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Yang Y, Parent J, Gil KM, Jones DJ. The Efficacy of Technology-Enhanced Behavioral Parent Training for Families With Low Income: Do Parent-Centered Profiles Moderate Treatment Outcomes? Behav Ther. 2025 Mar;56(2):261-275. doi: 10.1016/j.beth.2024.10.002. Epub 2024 Oct 18. PMID 40010899
- [Derived] Highlander A, Parent J, J Jones D. Helping the Noncompliant Child and Child Behavior Outcomes: An Exploratory Examination of Financial Strain. Prev Sci. 2025 May;26(4):542-554. doi: 10.1007/s11121-024-01749-9. Epub 2024 Nov 8. PMID 39514027
- [Derived] Parent J, Anton MT, Loiselle R, Highlander A, Breslend N, Forehand R, Hare M, Youngstrom JK, Jones DJ. A randomized controlled trial of technology-enhanced behavioral parent training: sustained parent skill use and child outcomes at follow-up. J Child Psychol Psychiatry. 2022 Sep;63(9):992-1001. doi: 10.1111/jcpp.13554. Epub 2021 Dec 9. PMID 34888861
- [Derived] Faro AL, McKee LG, Garcia RL, Jones DJ. The relationships between religiosity and youth internalizing symptoms in African American parent-adolescent dyads. Cultur Divers Ethnic Minor Psychol. 2018 Jan;24(1):139-149. doi: 10.1037/cdp0000158. Epub 2017 Jun 5. PMID 28581304
- [Derived] Anton MT, Jones DJ, Youngstrom EA. Socioeconomic status, parenting, and externalizing problems in African American single-mother homes: A person-oriented approach. J Fam Psychol. 2015 Jun;29(3):405-415. doi: 10.1037/fam0000086. PMID 26053349